CLINICAL TRIAL: NCT03010163
Title: Taxi STEP (Social Networks, Technology, and Exercise Through Pedometers)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 16-1659
Record Dates: First submitted 2017-01-03; First posted 2017-01-04 (Estimated); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Physical Conditioning
Keywords: pedometer; walking; taxi driver; 16-1659
MeSH Terms: conditions — Motor Activity | interventions — Health Fairs

ARMS (4):
- Health Fair + Pedometer (Active Comparator): Participants will get free weight, height, waist, and blood pressure testing at health fairs stationed at NYC taxi garage bases and airport taxi holding lots. Health fair staff will follow up with participants who need to see a doctor due to a high blood pressure reading or other unusual result that needs a physician follow-up. All participants will be given a pedometer with instructions on how to use it to track their daily step counts. Participants will be randomized by envelope provided by Memorial Sloan Kettering's Department of Epidemiology and Biostatistics during an in person meeting after the completion of the 1 month run-in or by phone in case we are unable to meet them in person.
  Interventions: Other: Health Fair; Other: Pedometer
- Health Fair, Pedometer + Text Messaging (Experimental): In addition to the health fair services with general follow-up, and giving each driver a pedometer with instructions on how to use the devise to track daily step counts, all participants in this group will receive daily healthy living advice and encouraging messages about walking through text messages sent by study staff to participants' cellular phone. Participants will be randomized by envelope provided by Memorial Sloan Kettering's Department of Epidemiology and Biostatistics during an in person meeting after the completion of the 1 month run-in or by phone in case we are unable to meet them in person.
  Interventions: Other: Health Fair; Other: Pedometer; Other: Text Messaging
- Health Fair, Pedometer, Social Network Support (Experimental): Each participant in this group will receive the health fair services with general follow-up along with a pedometer with instructions on how to use the device to track daily step counts. Additionally, participants in this group will be asked to provide the names of family or friends who will form a social support network team. This team will provide encouragement and remind participants to maintain a healthy lifestyle and increase daily walking activities. Participants will be given a social network guide to train their family and/or friends on how to best motivate the participants . Participants will be randomized by envelope provided by Memorial Sloan Kettering's Department of Epidemiology and Biostatistics during an in person meeting after the completion of the 1 month run-in or by phone in case we are unable to meet them in person.
  Interventions: Other: Health Fair; Other: Pedometer; Other: Social Network Support
- Health Fair, Pedometer, Text Msg, Social Network Support (Experimental): Participants in this group will receive the health fair service with general follow-up, along with a pedometer with instructions on how to use the device to track daily step counts. Participants will also receive daily healthy living advice through encouraging text messages about walking through text messages sent by our staff to participants' cellular phones. Participants will also be asked to provide the names of family or friends who will form a social support network team. This team will provide encouragement and remind participants to maintain a healthy lifestyle and increase daily walking activities. Participants will be given tools to train their family and/or friends on how to best motivate the drivers. Participants will be randomized by envelope provided by Memorial Sloan Kettering's Department of Epidemiology and Biostatistics during an in person meeting after the completion of the 1 month run-in or by phone in case we are unable to meet them in person.
  Interventions: Other: Health Fair; Other: Pedometer; Other: Text Messaging; Other: Social Network Support

INTERVENTIONS:
Other: Health Fair — Testing includes weight, height, waist and blood pressure testing. In the event that the participants are unable to meet in person for health measurements, the staff will accept self-reported measurements over the phone.
Other: Pedometer — The Fitbit One/Alta/Inspire wireless tracking pedometers measures steps taken, calories burned, distance traveled and sleep pattern. The Fitbit Alta/Inspire also sends reminders to move, which are notifications that remind the wearer to walk at least 250 steps each hour. If the wearer has not walked 250 steps within the hour, the device will vibrate and send an on-screen reminder 10 minutes before the hour. The reminders to move will be turned off during baseline and will be turned on at randomization for all participants.
Other: Text Messaging — Daily healthy living advice and encouraging messages about walking through text messages
  Arms: Health Fair, Pedometer + Text Messaging; Health Fair, Pedometer, Text Msg, Social Network Support
Other: Social Network Support — Family or friends will provide encouragement and remind participants to maintain in a healthy lifestyle and increase daily walking activities
  Arms: Health Fair, Pedometer, Social Network Support; Health Fair, Pedometer, Text Msg, Social Network Support

SUMMARY:
This study is divided into four groups. Group 1 includes Health Fairs implemented at NYC taxi garage bases and airport taxi holding lots and pedometers. Group 2 includes Health Fairs, pedometers and text messaging to facilitate walking and living a healthier lifestyle. Group 3 includes Health Fairs, pedometers and social network support. Group 4 includes Health Fairs, pedometers, text messaging and social network support.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Over 21 years of age
* Planning on remaining in NYC for at least 7 months
* Licensed taxi driver for at least three months
* Speaks English, Bengali, Hindi, Spanish or French
* Currently owns a cell phone, uses text messaging services and is willing to accept text messages for this study

Exclusion Criteria:

* Part-time driver (fewer than 5 shifts/week, totaling less than 35 hours per week)
* History of any CVD or any other medical conditions (e.g. severe osteoarthritis) that will prevent him from walking

  * Please note: All inclusion/exclusion criteria are based upon self reported information captured during study screening procedures.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2016-12; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Increase average daily step counts | 6 months post randomization
  Increase average step counts per day

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Gany, MD, MS, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

DOCUMENTS (1):
  • Informed Consent Form (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT03010163/ICF_000.pdf